CLINICAL TRIAL: NCT01976702
Title: Multi-Level HIV Prevention for Pregnant Drug Abusers
Acronym: PDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DESPR DA021521
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2013-10

CONDITIONS: Substance Related Disorders
Keywords: HIV risk behaviors; Pregnant drug abusers
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Behavioral Skills Training (Experimental): The Enhanced Behavioral Skills Training (E-BST) will include four 90-minute group sessions and two 60-minute individual sessions regarding HIV prevention and diminishing risk behavior, enhancing communication skills, improving the use of support services, and enhancing the use of resources in their community.
  Interventions: Behavioral: Enhanced Behavioral Skills Training
- Health Promotion Comparison (Active Comparator): The Health Promotion Comparison (HPC)condition will receive one video-based HIV prevention session, 3 video-based 90-minute group sessions and an additional 2 60-minute sessions with discussions on relevant topics unrelated to HIV.
  Interventions: Behavioral: Enhanced Behavioral Skills Training

INTERVENTIONS:
Behavioral: Enhanced Behavioral Skills Training

SUMMARY:
This 5 year study, targeting Pregnant Drug Abusers in treatment, is a randomized trial of an Enhanced Behavioral Skills Training (E-BST) intervention compared to a time-and attention-matched Health Promotion Comparison (HPC) condition. E-BST is an adaptation of the original BST intervention (Eldridge, St. Lawrence et al., 1997), designed to strengthen relationship-based social competency skills of the original BST that were crucial in sustaining adherence to protective behavior.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* a recent history (within the past year) of using illicit substances
* 12-32 weeks pregnant and not planning to terminate the pregnancy
* able to read English Informed Consent form; understand and provided written informed consent
* have competency in conversational English which is required to complete assessments and to participate in the intervention groups
* have a stable living arrangement and provide contact information
* currently not cognitively impaired since cognitive impairment may compromise the ability to comprehend and participate in the assessment and intervention
* currently not showing symptoms of a major psychiatric disorder/ including psychosis, or a high risk for suicidality
* report at least one episode of unprotected vaginal/anal sex since becoming pregnant
* answer "Yes" to this question: "Do you plan to be in the area for the next 12 months?"
* agree to a urine test at the time of each interview to detect the presence of drugs

Exclusion Criteria:

* under age 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2006-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Sexual risk behavior | 6 months post intervention
  Reduction in HIV sex risk and drug abuse behavior among pregnant substance abusers

SECONDARY OUTCOMES:
Drug use risk behavior | 6 months post intervention

OTHER OUTCOMES:
Service utilization, social support, and individual cognitive-behavioral factors | 6 months post intervention